CLINICAL TRIAL: NCT04838964
Title: An Open-label, Single-arm, Multi-center, Phase II Clinical Study of MRG003 in the Treatment of Patients With EGFR-positive Unresectable, Locally Advanced or Metastatic Biliary Tract Cancer
Brief Title: A Study of MRG003 in the Treatment of EGFR-positive Unresectable, Locally Advanced or Metastatic Biliary Tract Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Miracogen Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MRG003-003
Record Dates: First submitted 2021-04-06; First posted 2021-04-09 (Actual); Last update posted 2021-12-29 (Actual); Status verified 2021-12

CONDITIONS: Advanced or Metastatic Biliary Tract Cancer
Keywords: MRG003; Antibody Drug Conjugate (ADC); EGFR; Biliary Tract Cancer
MeSH Terms: conditions — Biliary Tract Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MRG003 (Experimental): MRG003 will be administrated via IV infusion at 2.0 mg/kg on Day 1 of every 3 weeks (21-day cycle).
  Interventions: Drug: MRG003

INTERVENTIONS:
Drug: MRG003 — Administrated intravenously

SUMMARY:
The objective of this study is to assess the safety, efficacy, pharmacokinetics, and immunogenicity of MRG003 as single agent in EGFR-positive unresectable locally advanced or metastatic biliary tract cancer patients who have progressed during or relapsed after at least one prior standard therapy.

DETAILED DESCRIPTION:
The study consists of two stages. In Phase IIa, approximately 25 subjects will be enrolled to evaluate the safety and preliminarily efficacy of MRG003. Based on the safety and efficacy data obtained from the Phase IIa, the study design of the second stage Phase IIb single-arm study either will be adjusted or the trial will be stopped. If the initial Phase IIa data support the continuation of the study, in the second stage, approximately an additional 55 subjects will be enrolled to further evaluate the efficacy and safety of MRG003.

ELIGIBILITY:
Inclusion Criteria:

1. Willing to sign the ICF and follow the requirements specified in the protocol.
2. Aged 18 to 75 (including 18 and 75), both genders.
3. Expected survival time ≥ 12 weeks.
4. Patients with unresectable locally advanced or metastatic biliary tract cancer confirmed by histopathology.
5. Failed in the prior one or more standard therapies.
6. EGFR positive in the tumor specimens confirmed by central laboratory test.
7. Archival or biopsy tumor specimens should be provided (primary or metastatic).
8. Patients must have measurable lesions according to the Response Evaluation Criteria in Solid Tumors (RECIST v1.1).
9. ECOG performance score 0 or 1.
10. Prior anti-tumor treatment-related AEs (NCI CTCAE v5.0 Criteria) have recovered to ≤ Grade 1 (except alopecia, non-clinically significant or asymptomatic laboratory abnormalities).
11. No severe cardiac dysfunction with left ventricular ejection fraction (LVEF) ≥ 50%.
12. Organ function must meet the basic requirements.
13. Coagulation function must meet the basic requirements.
14. Patients of childbearing potential must take effective contraceptive measures during the treatment and for 6 months after the last dose of treatment.

Exclusion Criteria:

1. History of hypersensitivity to any component of MRG003.
2. Received chemotherapy, radiotherapy, biologicals, immunotherapy, or other anti-tumor drugs within 4 weeks prior to the first dose.
3. Presence of clinical manifestation of biliary obstruction.
4. Patients with clinical symptoms such as pleural, abdominal or pericardial effusion requiring puncture drainage.
5. Presence of central nervous system (CNS) metastasis and/or neoplastic meningitis.
6. Any severe or uncontrolled systemic diseases.
7. Patients with poorly controlled heart diseases.
8. Evidence of active infections, including but not limited to Hepatitis B, Hepatitis C, or human immunodeficiency virus (HIV) infection.
9. History of other primary malignancies.
10. History of the following ophthalmologic abnormalities：severe dry eye syndrome; keratoconjunctivitis sicca; severe exposure keratitis; any other condition that may increase the risk of corneal epithelial damage.
11. History of severe skin disease or chronic skin disease requiring oral or intravenous treatment.
12. History of interstitial pneumonia, severe chronic obstructive pulmonary disease, severe pulmonary insufficiency, symptomatic bronchospasm, etc.
13. Peripheral neuropathy greater than Grade 1.
14. Patients with active autoimmune disease or a history of autoimmune disease, who are using immunosuppressive agents, or systemic hormone therapy and still receiving within 2 weeks prior to enrollment.
15. History of cirrhosis (decompensated cirrhosis Child-Pugh class B and C).
16. Received anti-tumor vaccine treatment 4 weeks prior to the first dose or planning to participate in anti-tumor vaccine trials.
17. Female patents with a positive serum pregnancy test or who are breast-feeding or who do not agree to take adequate contraceptive measures during the treatment and for 6 months after the last dose of study treatment.
18. Other conditions inappropriate for participation in this clinical trial, at the discretion of the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-04-28 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) by Independent Review Committee (IRC) | Baseline to study completion, up to 12 months
  ORR is defined as the percentage of patients with a complete response (CR) and partial response (PR) as assessed by Independent Review Committee (IRC) according to RECIST v1.1.

SECONDARY OUTCOMES:
ORR by Investigator | Baseline to study completion, up to 12 months
  ORR is defined as the percentage of patients with a CR and PR as assessed by Investigator according to RECIST v1.1.
Duration of Response (DoR) | Baseline to study completion, up to 12 months
  DOR is defined as the time from first documented objective response to the first onset of tumor progression or death of any cause.
Time to Response (TTR) | Baseline to study completion, up to 12 months
  TTR is defined as the duration from the start of treatment to the first onset of CR or PR in tumor evaluation.
Disease Control Rate (DCR) | Baseline to study completion, up to 12 months
  DCR is defined as the percentage of patients who achieve CR, PR, and stable disease (SD) after treatment.
Progression Free Survival (PFS) | Baseline to study completion, up to 12 months
  PFS is defined as the duration from the start of treatment to the onset of tumor progression or death of any cause.
Overall Survival (OS) | Baseline to study completion, up to 12 months
  OS is defined as the duration from the start of treatment to death of any cause.
Adverse Events (AEs) | Baseline to 30 days after the last dose of study treatment
  Any reaction, side effect, or untoward event that occurs during the course of the clinical trial whether or not the event is considered related to the study drug.
Pharmacokinetics (PK) parameter of MRG003: concentration-time curve | Baseline to 30 days after the last dose of study treatment
  Concentration-time curve will be depicted based on pharmacokinetics concentration set (PKCS).
Incidence of anti-drug antibody (ADA) | Baseline to 30 days after the last dose of study treatment
  The incidence of ADA analysis will be summarized for all patients who received at least one cycle study treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Aiping Zhou, MD, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (7):
- China (7):
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Beijing Youan Hospital,Capital Medical University, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Hunan Cancer Hospital, Changsha, Hunan
  - Bethune First Hospital of Jilin University, Changchun, Jilin

IPD SHARING:
Plan to Share IPD: No